CLINICAL TRIAL: NCT03091959
Title: Profiling of Implantable Cardiac Device Diagnostics Trends During Clinical Events for Co-morbid Conditions in Indian Patients- PATTERNS Study
Brief Title: Profiling Implantable Cardiac Device Diagnostics Trends During Clinical Events .
Acronym: PATTERNS
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16044
Record Dates: First submitted 2017-02-24; First posted 2017-03-27 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study looks to evaluate the device diagnostic data obtained from (all the Cardiac Rhythm and Heart Failure (CRHF) devices of medtronic having the Cardiac Compass® and OptiVol® diagnostic feature) these devices to identify trends during clinical events that will help early detection and prevention of cardiovascular and other comorbid conditions. (i.e. Heart failure(HF), Atrial Fibrilation,COPD, Renal dysfunction (RD), Diabetes etc.)

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, Non-interventional, data collection study with no subject follow-up visits required. Subjects will be enrolled and exited from the study during the same study visit.

The final analysis on the study will occur when 50 clinical events are reported on the study.All Medtronic implantable Cardiac Rhythm and Heart Failure devices with the Cardiac Compass® and OptiVol® feature which are commercially available at the start of the registry or become commercially available during the course of the registry and used within its intended use, may be included in the study.

After obtaining the informed consent patients will be interviewed to complete the "patient interview questionnaire". The study team will review medical records and complete the "Medical Record Review" form as completely as possible. The device will then be interrogated to download the cardiac Compass® report in a "save-to-disk" file and print the cardiac Compass® report for the PI or the designated clinician from the study team for review. The "device interrogation questionnaire" will then be discussed with the patient for specific events identified on the Cardiac Compass® report in order to determine possible explanations and fill out the questionnaire as completely as possible. After collection of all the study related data the patient will be exited on the same visit, so a followup visit is not required in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be greater than 18 years of age.
2. Subject must have an implanted Medtronic CRHF device (with the Optivol® and Cardiac Compass® diagnostics) for at least 1 year.
3. Subjects between 18 years and 62 years of age must have at least 1 clinical event ,such as any major medication change, IV drug therapy, hospitalization, outside home-treatment or any similar event in the past 1 year from the date of enrollment which required a Pharmacologic intervention, associated with any of the following comorbid conditions :

   * Heart failure
   * Chronic Obstructive Pulmonary Disease (COPD)
   * Renal deficiency
   * Atrial fibrillation
   * Diabetes
4. Subjects who are currently hospitalized with an Index clinical event can also be enrolled.
5. If the subject is over 62 years of age then subject can be enrolled in the study without any pre-condition of a clinical event associated with a comorbid condition.

Exclusion Criteria:

* Subject is unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 300 subjects (i.e. consented) from upto 7 sites. All subjects implanted with devices (Medtronic Cardiac Rythm and Heart Failure (CRHF) implantable devices with Cardiac compass and Optivol feature) will be considered eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in device measured diagnostic parameters | The diagnostic parameters can be stored within device for upto 12 months and this will be evaluated once the patient is interrogated and the report analyzed.
  Determine a combined diagnostic index that can identify patient at risk for a clinical event Determine the number of device measured diagnostic parameter that change prior to any clinical events associated with at least one of the comorbid conditions, including worsening heart failure, COPD, diabetes, and renal failure, which require major medication change, IV drug therapy, hospitalization, outside home treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Rajan, Phd, Study Chair — Medtronic
Locations (4):
- India (4):
  - Medanta - The Medicity, Gurgaon, Haryana
  - LISIE Hospital, Kochi, Kerala
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Escort Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No
All patient identifiers will be anonymized and only the final results will be shared if there is a need.

REFERENCES:
- [Background] Prabhakaran D, Jeemon P, Roy A. Cardiovascular Diseases in India: Current Epidemiology and Future Directions. Circulation. 2016 Apr 19;133(16):1605-20. doi: 10.1161/CIRCULATIONAHA.114.008729. PMID 27142605
- [Background] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Circulation. 2003 Oct 28;108(17):2154-69. doi: 10.1161/01.CIR.0000095676.90936.80. No abstract available. PMID 14581387
- [Background] Tharkar S, Satyavani K, Viswanathan V. Cost of medical care among type 2 diabetic patients with a co-morbid condition--hypertension in India. Diabetes Res Clin Pract. 2009 Feb;83(2):263-7. doi: 10.1016/j.diabres.2008.11.027. Epub 2008 Dec 31. PMID 19118912
- [Background] Varma PP. Prevalence of chronic kidney disease in India - Where are we heading? Indian J Nephrol. 2015 May-Jun;25(3):133-5. No abstract available. PMID 26060360
- [Background] Vijayan VK. Chronic obstructive pulmonary disease. Indian J Med Res. 2013 Feb;137(2):251-69. PMID 23563369
- [Background] Chhabra SK, Gupta M. Coexistent chronic obstructive pulmonary disease-heart failure: mechanisms, diagnostic and therapeutic dilemmas. Indian J Chest Dis Allied Sci. 2010 Oct-Dec;52(4):225-38. PMID 21302600